CLINICAL TRIAL: NCT00407342
Title: Prospective, Randomized Half-side Comparison of Alefacept (Amevive) With or Without UVB-311nm Phototherapy in Patients With Psoriasis (Translated From German)
Brief Title: Alefacept (Amevive) With or Without Narrowband UVB Treatment in Patients With Psoriasis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Peter Wolf, MD, Principal Investigator, Medical University of Graz, Austria
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-075ex03/04
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Psoriasis
Keywords: Psoriasis; biologics; alefacept; Narrowband UVB; Phototherapy; Half-side comparison
MeSH Terms: conditions — Psoriasis | interventions — Alefacept; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alefacept (drug) — alefaceptgiven iv
  Other Names: Amevive
Procedure: Narrowband UVB phototherapy

SUMMARY:
Alefacept is a new anti-psoriatic drug within the group of the so-called biologics. In about 30% of patients alefacept induces a more than 75% improvement of psoriasis after a 12-week treatment period. The start of anti-psoriatic effect by alefacept is delayed, however improvement of psoriatic lesions outlasts the end of alefacept treatment.

Narrowband UVB (UVB-311nm) phototherapy is an established anti-psoriatic treatment regimen with rapid onset of anti-psoriatic efficacy but disease-free intervals after the end of successful treatment courses may be short.

Therefore, in this half-side (left/right side) comparison study we aim to investigate whether an additional narrowband UVB treatment accelerates and improves the anti-psoriatic treatment effects of alefacept.

DETAILED DESCRIPTION:
Psoriasis is an inflammatory skin disease that affects an estimated 2% to 3% of the world's population. There are a wide range of local and systemic clinical treatments and agents for clearing, or at least reducing the expression of, psoriatic skin lesions. There is a new generation of antipsoriatic drugs that specifically target T-cell mediated inflammatory pathways and that are approved for the treatment of moderate to severe psoriasis in the United States. Alefacept (Amevive) is one of these so-called biologics. Alefacept appears to have several advantages over other systemic antipsoriatic agents and is very well tolerated by patients. Weekly administration of alefacept for 12 weeks reduced the psoriasis area and severity index (PASI) by greater than 75% in 30% of patients. The maximal antipsoriatic effect, however, apparently occurs after the 12-week course has ended. In vitro studies and previous case reports suggested that alefacept's antipsoriatic effect may be augmented when it is administered in combination with UVB. These findings prompted us to conduct a prospective randomized half-body comparison study, in which we ask whether the clinical response of psoriatic lesions to alefacept could be improved by combining alefacept with standard UVB 311nm phototherapy.

Comparison: Psoriatic patients are treated with intravenous alefacept once per week for 12 weeks. One randomized chosen body-half (left or right side) is additionally treated with narrowband UVB (UVB-311nm) three times per week until complete clearance of psoriatic lesions at the UV-treated side. PASI is evaluated before, weekly during, and for 3 to 12 months after alefacept +/- narrowband UVB treatment.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe plaque-type psoriasis;
* disease duration for more than 6 months
* PASI above 10.

Exclusion Criteria:

* age < 18 years;
* pregnancy or lactation;
* presence of a dysplastic nevus syndrome;
* photosensitive skin disease;
* autoimmune disease;
* severe renal or hepatic disease;
* presence or history of malignant skin tumors;
* presence of antinuclear antibodies;
* history of previous treatments with arsenic, methotrexate, or x-rays;
* within the last 4 weeks before enrollment into the study, UVB or PUVA treatment, immunosuppressive/-modulating drugs (such as corticosteroids, cyclosporine, and biologics such as infliximab, etanercept or efalizumab).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-02; Primary Completion 2004-06 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Modified PASI (Psoriasis area and severity index) | 6 months

SECONDARY OUTCOMES:
VAS for therapeutic effect; | 6 months
VAS for severity of skin lesions | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Research Unit for Photodermatology, Department of Dermatology, Medical University Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

REFERENCES:
- [Derived] Legat FJ, Hofer A, Wackernagel A, Salmhofer W, Quehenberger F, Kerl H, Wolf P. Narrowband UV-B phototherapy, alefacept, and clearance of psoriasis. Arch Dermatol. 2007 Aug;143(8):1016-22. doi: 10.1001/archderm.143.8.1016. PMID 17709660